CLINICAL TRIAL: NCT01505959
Title: Blood Pressure Reduction Induced by Continuous Positive Airway Pressure (CPAP) in Sleep Apnea Patients at High Cardiovascular Risk : A Randomized Controlled Trial Comparing Usual CPAP Care Versus a Multidisciplinary and Coordinated Follow-up Based on a Telemonitoring Web Platform
Brief Title: Blood Pressure Reduction Induced by CPAP in Sleep Apnea Patients at High Cardiovascular Risk : OPTISAS 2 Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fédération Française de Pneumologie (Other)
Collaborators: Federation of Medical Specialties (Other)
Responsible Party: Principal Investigator, Jean Louis PEPIN, Professor, PhD, Hospital Grenoble France, Fédération Française de Pneumologie
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-FFPO-02
Record Dates: First submitted 2012-01-05; First posted 2012-01-09 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Sleep Apnea Syndromes; High Cardiovascular Risk
Keywords: Obstructive Sleep Apnea Syndrome; Apnea; Sleep Apnea; Telemedicine; CPAP compliance
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Apnea | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional (Experimental)
  Interventions: Device: CPAP treatment
- Telemedicine (Active Comparator)
  Interventions: Device: CPAP treatment

INTERVENTIONS:
Device: CPAP treatment — Usual CPAP treatment
  Arms: Conventional
Device: CPAP treatment — CPAP treatment with telemedicine system
  Arms: Telemedicine

SUMMARY:
Targeted population:

Sleep apnea patients at high cardiovascular risk newly treated by CPAP

Hypothesis:

Improvement in blood pressure after 6 months of CPAP treatment might be greater in the telemonitoring arm compared to usual CPAP care.

Main goal:

To compare 6-months blood pressure reduction when Sleep Apnea patients at high cardiovascular risk are randomly allocated to usual CPAP care or a multidisciplinary and coordinated follow-up based on a telemonitoring web platform.

DETAILED DESCRIPTION:
Study procedures:

The telemonitoring system will involve respiratory physicians, home care providers and include regular assessments of home self-measured blood pressure, oximetry, physical activity recorded by actigraphy, CPAP compliance, side effects and residual events.

Secured data transmission to medical staff computers and secured websites will allow easy telemonitoring. Automatic algorithms have been built-up for early adjustment of CPAP treatment in case of side effects, leaks and persistent residual events.

An interim analysis will be performed when 300 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 78 years
* Men and women
* AHI > 30 / hour
* Patient with high cardiovascular score (>5% defined by European SCORE) or known cardiovascular disease (i.e. transient ischemic attack, stroke, coronary artery disease)
* Patient affiliated to the National health insurance
* Willingness to use a telemonitoring system

Exclusion Criteria:

* Central sleep apnea syndrome
* Previous CPAP treatment with respiratory support for sleep respiratory trouble
* Cardiac failure with left ventricular ejection fraction lesser than 40%
* Hypercapnic chronic respiratory failure (daytime PaCO2 > 50 mmHg)
* Terminal disease

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 936 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure evolution by comparing baseline and 6 months measurements | day 0 and month 6
  Systolic blood pressure is assessed at day 0 and month 6 in the two groups by home self-measured blood pressure (4 consecutive days)

SECONDARY OUTCOMES:
Objective CPAP compliance at 6 months | day 0 and month 6
  CPAP compliance assessed after 6 months in the two groups
Diastolic blood pressure evolution by comparing baseline and 6 months | day 0 and month 6
  Diastolic blood pressure is assessed at day 0 and month 6 in the two groups
Subjective Sleepiness | inclusion and month 6
  Sleepiness is assessed with Epworth Sleepiness Scale at inclusion and month 6 in the two groups
Fatigue | inclusion and month 6
  Fatigue is assessed with Pichot Scale at inclusion and month 6 in the two groups
Quality of Life | inclusion and month 6
  Quality of life is assessed with SF-12 questionnaire at inclusion and month 6 in the two groups
Health status | inclusion and month 6
  Health status is assessed with EQ-5D questionnaire at inclusion and month 6 in the two groups
Physical activity | inclusion and month 6
  Physical activity is assessed with actimetry at inclusion and month 6 in the two groups
Cost analysis | month 6
  Cost analysis will include all key resources associated with the telemonitoring intervention and related health (referrals, consultations, resource use)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis PEPIN, Prof, PhD, Principal Investigator — University Hospital, Grenoble, France
Locations (32):
- France (32):
  - Respiratory physician in private practice, Albertville
  - Respiratory physician in private practice, Annecy
  - Respiratory physician in private practice, Bordeaux
  - General Hospital, Cannes
  - General Hospital, Denain
  - Dieulefit Santé Clinic, Dieulefit
  - Respiratory physician in private practice, Échirolles
  - Saint Vincent Clinic, Épernay
  - Respiratory physician in private practice, Grenoble
  - University Hospital, Grenoble
  - Respiratory physician in private practice, La Rochelle
  - University Hospital Calmette, Lille
  - La Louvière Clinic, Lille
  - General Hospital, Magny-en-Vexin
  - Ambroise Paré Hospital, Marseille
  - General Hospital, Montélimar
  - Respiratory physician in private practice, Montigny-lès-Metz
  - Respiratory physician in private practice, Nîmes
  - Les Rieux Clinic, Nyons
  - Hospital Bichat Claude Bernard, Paris
  - Respiratory physician in private practice, Reims
  - University Hospital, Rouen
  - General Hospital, Saint-Avold
  - Respiratory physician in private practice, Saint-Etienne
  - Respiratory physician in private practice, Saint-Ismier
  - Respiratory physician in private practice, Saint-Laurent-du-Var
  - Respiratory physician in private practice, Saint-Omer
  - Respiratory physician in private practice, Six-Fours-les-Plages
  - Respiratory physician in private practice, Toulon
  - Respiratory physician in private practice, Valence
  - Tessier Clinic, Valenciennes
  - Hospital Nord Ouest, Villefranche-sur-Saône